CLINICAL TRIAL: NCT01672931
Title: The Association Between Overweight and Oocyte Diameter in Women Undergoing Vitro Fertilization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0034-12 HYMC
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Infertility; Obesity
MeSH Terms: conditions — Infertility; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BMI over 30: Women undergoing IVF with BMI over 30
  Interventions: Other: Oocyte Measurement
- BMI 20-25: Women undergoing IVF treatments with BMI between 20-25
  Interventions: Other: Oocyte Measurement

INTERVENTIONS:
Other: Oocyte Measurement

SUMMARY:
We believe that there is an association between BMI and oocyte diameter in women undergoing IVF treatments. We plan to measure the oocyte diameter in 2 groups of women undergoing IVF. One group will have BMI 20-25 and the other group will have BMI above 30.

ELIGIBILITY:
Inclusion Criteria:

* IVF treated patients
* BMI between 20-25 or over 30

Exclusion Criteria:

* Everyone else

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing IVF treatments
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Larger Size of Oocyte Diameter | One year
  Oocyte will be measured in women undergoing IVF treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gai Shrem, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] Atzmon Y, Shoshan-Karchovsky E, Michaeli M, Aslih N, Shrem G, Ellenbogen A, Shalom-Paz E. Obesity results with smaller oocyte in in vitro fertilization/intracytoplasmic sperm injection cycles-a prospective study. J Assist Reprod Genet. 2017 Sep;34(9):1145-1151. doi: 10.1007/s10815-017-0975-6. Epub 2017 Jun 17. PMID 28624860